CLINICAL TRIAL: NCT04151394
Title: Side-to-side Duodenojejunostomy After Resection of Third and Fourth Duodenal Part With Pancreatic Preservation
Brief Title: Side-to-side Duodenojejunostomy After Distal Duodenal Resection (DUORESECT)
Acronym: DUORESECT
Status: Completed | Type: Observational
Sponsor: Universidad de Extremadura (Other)
Collaborators: Complejo Hospitalario Universitario de Badajoz (Other)
Responsible Party: Principal Investigator, Gerardo Blanco-Fernández, Head of Surgery, Clinical Professor, Universidad de Extremadura
Other Study IDs: UE-CHUB 001-2019
Record Dates: First submitted 2019-10-31; First posted 2019-11-05 (Actual); Last update posted 2019-11-18 (Actual); Status verified 2019-11

CONDITIONS: Duodenal Neoplasm; Gastrointestinal Disease; Surgery--Complications; Survival
MeSH Terms: conditions — Duodenal Neoplasms; Gastrointestinal Diseases

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 12 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Duodenojejunostomy — Resection of duodenal lesions and reconstruction by duodenojejunostomy

SUMMARY:
Lower partial duodenectomy could be indicated in case of injury, wide neck diverticulum, tumor invasion by other tumors such as retroperitoneal sarcoma and primary tumor of 3rd and 4th portion of the duodenum. Reconstruction after resection is usually performed by a end-to-end or end-to-side anastomosis.

The investigators analyze the short and long-term results of a case series with resection for various lesions in the third and fourth duodenal portions and reconstruction of the intestinal transit through side-to-side duodenojejunostomy

DETAILED DESCRIPTION:
The investigators retrospectively looked at patients who, from January 2010 to December 2018, underwent surgical procedures for duodenal tumors or other type of primary lesions.

Patients with primary duodenal lesions who underwent surgery were included in the study. Patients with secondary duodenal infiltration or liver and/or peritoneal metastasis found during intraoperative exploration were excluded. Similarly, if the surgeons appreciate the involvement of the pancreas during the procedure, for which they would have to perform a pancreaticoduodenectomy, the patient would be excluded.

Diagnostic management included establishment of a medical history, performance of clinical examination and imaging tests, including endoscopic exploration and, when neoplasm was suspected, computerized tomography (CT) scan, to confirm the tumor origin and growth, as well as infiltration, if any, of adjacent structures. These also allowed to rule out distant metastases, and to assess resectability and the option for reconstruction according to the location.

The variables taken into account were age, sex, the American Society of Anesthesiologists (ASA) classification, preoperative examinations performed and type of lesion susppected as benign, duodenal adenocarcinoma or gastrointestinal stromal tumor (GIST). Perioperative clinical results, surgical approach, type of resection and reconstruction, and intraoperative complications were recorded. Details of the postoperative course were collected. Some of the key short-term data recorded included length of hospital stay, complications' ranking (according to the Clavien-Dindo score; 'severe complication' is defined as greater or equal to IIIa), re-operation, re-admission and operative mortality (< 90 days after operation). Some of the key long-term data recorded were, digestive symptoms along follow-up, specific disease-free survival (DFS) and overall survival (OS)

ELIGIBILITY:
Inclusion Criteria:

* Patients with primary duodenal lesions who underwent surgery

Exclusion Criteria:

* Secondary duodenal infiltration or liver and/or peritoneal metastasis found during intraoperative exploration

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who, from January 2010 to December 2018, underwent surgical procedures in our unit for duodenal tumors or other type of primary lesions.
Sampling Method: Non-Probability Sample
Enrollment: 13 (Actual)
Dates: Start 2019-01-31 (Actual); Primary Completion 2019-09-01 (Actual); Study Completion 2019-10-01 (Actual)

PRIMARY OUTCOMES:
Complication | 90 days
  Surgical complications rates
Overall survival | 10 years
  Patients overall survival after resection

CONTACTS AND LOCATIONS:
Locations (1):
- Gerardo Blanco-Fernández, Badajoz, Spain

IPD SHARING:
Plan to Share IPD: Undecided